CLINICAL TRIAL: NCT00988702
Title: Shaolin Dan Tian Breathing Fosters Relaxed and Attentive Mind: A Randomized Controlled Neuroelectrophysiological Study
Brief Title: Shaolin Dan Tian Breathing Fosters Relaxed and Attentive Mind
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Chinese University of Hong Kong (Other)
Responsible Party: Dr. Mei-chun Cheung, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: Chanwuyi-0006
Record Dates: First submitted 2009-09-30; First posted 2009-10-02 (Estimated); Last update posted 2009-10-02 (Estimated); Status verified 2009-10

CONDITIONS: Attention; Electroencephalography
Keywords: Dan Tian Breathing; Physiological measurement; progressive muscle relaxation; Monitoring, Physiologic
MeSH Terms: interventions — Autogenic Training

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dan Tian Breathing (Experimental): subjects received one-month's training on the Dan Tian Breathing
  Interventions: Behavioral: Dan Tian Breathing
- Progressive muscle relaxation training (Active Comparator): Subjects received one-month's conventional progressive muscle relaxation training
  Interventions: Behavioral: Progressive muscle training

INTERVENTIONS:
Behavioral: Dan Tian Breathing — Dan Tian Breathing for one month
  Other Names: Dan Tian; Shaolin
  Arms: Dan Tian Breathing
Behavioral: Progressive muscle training — Progressive muscle training for one month
  Other Names: muscle training; relaxation
  Arms: Progressive muscle relaxation training

SUMMARY:
The present study aimed to utilize these well-known neuroelectrophysiological techniques to investigate the relatively less studied Shaolin Dan Tian Breathing (DTB) technique.

DETAILED DESCRIPTION:
Neuroelectrophysiological studies on various types of meditative breathing revealed its association with either a relaxing (i.e., enhanced alpha asymmetry) or an attentive state (i.e., enhanced intra- and inter-hemispheric theta coherence). The present study aimed to utilize these well-known neuroelectrophysiological techniques to investigate the relatively less studied Shaolin Dan Tian Breathing (DTB) technique. This technique consists of two components -- Passive DTB and Active DTB, and is considered not only as a relaxation exercise but also a form of Qigong. Based upon some pilot neuroimaging data and clinical observation, it was hypothesized that after familiarizing with the method, practicing DTB can induce both relaxing and attentive states. Twenty-two adults received training on the DTB (experimental group) for one month. They were instructed to practice the technique daily, and at each practice, until they felt warm and/or relaxed. Twenty age-, gender- and education-matched adults receiving conventional progressive muscle relaxation training were recruited as control. All participation was voluntary. Quantitative EEG and bio-physiological data were collected at baseline and post training. Eyes-closed resting EEG data before and immediately after each type of breathing were obtained individually at two time points.

ELIGIBILITY:
Inclusion Criteria:

* healthy controls
* age 20 to 60 years

Exclusion Criteria:

* history of head injury,
* seizure,
* stroke,
* other CNS diseases or psychiatric illnesses of psychosis or mania.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2008-10; Primary Completion 2009-03 (Actual); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Quantitative electroencephalography | Before and after one month's training

SECONDARY OUTCOMES:
Bio-physiological measures | Before and after one month's training

CONTACTS AND LOCATIONS:
Overall Officials: Agnes S Chan, PhD, Principal Investigator — The ChineseUniversity of Hong Kong